CLINICAL TRIAL: NCT00001247
Title: Inpatient Evaluation of Neuropsychiatric Patients
Brief Title: Inpatient Evaluation of Adults With Schizophrenia
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 890160; 89-M-0160
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-04-18

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Psychosis; Schizoaffective; Neuroimaging; Cognition; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Sirolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Individuals with schizophrenia-spectrum illness from the community.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Drug not used in study.

SUMMARY:
The purpose of this study is to understand the biologic basis of schizophrenia and to determine which symptoms are related to the illness itself and which are related to medications used to treat the illness.

Schizophrenia and related psychoses are chronic brain disorders whose prognosis is often poor and whose pathophysiology remains obscure. Brain imaging technologies such s positron emission tomography (PET), functional magnetic resonance imaging (fMRI), and magnetic resonance imaging (MRI) offer opportunities to study the pathophysiology of psychotic disorders by evaluating brain function. However, the use of anti-psychotic drugs may interfere with the results of such studies. In this study, psychotropic medication will be discontinued in patients for a short period of time to distinguish the effects of the illness on the brain without the interference of the medication's effects on the brain. Given that there is a risk that the patient's symptoms will increase, they are asked to stay on an inpatient unit where the NIMH clinical staff is available to help them 24 hours a day.

This study will be conducted in three phases. In Phase 1, participants will be admitted to the Clinical Center while continuing to take their medication and will undergo diagnostic interviews, physical and laboratory assessments, physiological monitoring, and neuropsychological testing. Behavioral ratings will also be performed and blood and urine samples will be collected. During Phase 2, participants will continue taking medications in a blinded fashion for 8 to 12 weeks. The active medications will be replaced with a placebo (an inactive pill) part of that time. PET, fMRI, and MRI scans will be used to monitor how the continuation or lack of medication affects the brain. Psychological tests will also be given to measure changes in cognition. In Phase 3, participants will have the opportunity for clinical stabilization.

DETAILED DESCRIPTION:
Objectives:

Schizophrenia and related psychoses are chronic brain disorders whose prognosis is often poor and whose pathophysiology remains obscure. Neuroimaging technologies such as PET (positron emission tomography), fMRI (functional magnetic resonance imaging), DTI (diffusion tensor imaging) and MRSI (magnetic resonance spectroscopic imaging) offer opportunities to elucidate the pathophysiology by studying brain function in living research subjects. The use of these techniques to study psychotic disorders is severely limited, however, by a critical methodological confound: antipsychotic treatment. The purpose of this protocol is to admit research subjects with schizophrenia and other related disorders to the Clinical Center, carefully evaluate their neuropsychiatric status, and discontinue psychotropic medications for a brief period so research subjects can be studied without the confound of antipsychotic treatment.

Study Population:

700 participants

The study will include research subjects with schizophrenia.

Study Design:

There are several phases to this protocol. The first phase is the Screening Evaluation and Stabilization Phase and includes gathering historical data, structured diagnostic interviews, general physical and laboratory assessments, basic physiological monitoring, neuropsychological testing, limited collection of blood and urine samples, and serial behavioral ratings. In the second phase (Coded Medication Phase), research subjects will receive blinded compounds that will contain inactive placebo or active antipsychotic administered in a crossover fashion. Patients and unit clinical nursing staff evaluating and caring for the patient will be blind to arm status. Each arm normally lasts 4 to 6 weeks. The total duration of this phase is 8 to 12 weeks. During the Coded Medication Phase, research subjects are enrolled in a series of neuroimaging and other approved studies designed to elucidate the neurobiology of these disorders. These include studies using neuropsychological testing, MEG, PET, fMRI, DTI, and MRSI. The antipsychotic free period is essential to distinguish the effects of illness versus medication.

Outcome Measures:

Parameters under investigation include traits that are candidate phenotypes for genetic studies and state-dependent aspects of brain function. The combined use of many neuroimaging modalities will allow us to look at the functional relationship between a variety of brain abnormalities hypothesized to play a role in schizophrenia. These include hippocampal neurochemical abnormalities, deficits in prefrontal cortical activation, and dysregulation of subcortical dopamine in a single research subject.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Diagnosis of DSM-IV- or DSM5-defined schizophrenia spectrum disorder (including schizophrenia, schizoaffective disorder, or other specified/unspecified schizophrenia spectrum and other psychotic disorder/psychosis NOS).

Subjects with other neuropsychiatric disorders may also be admitted and participate in the protocol if there is sufficient evidence to believe they have an underlying, undiagnosed DSM-IV-or DSM5-defined schizophrenia spectrum disorder.

EXCLUSION CRITERIA:

-Currently treated with depot medications

Because of the long half-life of depot medications such as paliperidone palmitate (Invega Sustenna), applicants to our program will be excluded if they are currently receiving depot medications monthly. However, applicants may decide to switch from depot to oral medications on their own, in conjunction with their personal physician, before coming to the program. This is not part of research and we do not participate in this decision. A sufficient washout period based on the particular long-acting injectable medication s elimination half-life will be required in order for prospective participants to be eligible. Subjects may complete the last 3 months of washout in the inpatient unit while being evaluated under the standard protocol.

-Major medical illness.

Research subjects identified as having major medical problems other than their primary neuropsychiatric disorder will be excluded from admission.

* Applicants judged to be unsuitable for medication free studies will also be excluded. Possible reasons for exclusion include prior history of dangerousness to self or others, particularly when off medication.
* Applicants who are pregnant are excluded from this study. Volunteers who are found to be pregnant after testing will be terminated from study and referred to an OB-GYN for follow up care.
* Infection with syphilis, hepatitis, or HIV.
* History of any (excepting nicotine-related and cannabis-related) DSM5-defined moderate to severe substance use disorder (or DSM-IV-defined substance dependence).
* Cumulative lifetime history of any (excepting nicotine-related and cannabis-related) DSM5-defined mild substance use disorder (or any DSM-IV-defined substance abuse), either in excess of 5 years total or not in remission for at least 6 months.
* Lack of capacity to provide consent.

Exclusion Criteria for Previously Enrolled Research Subjects

* No longer satisfying the above inclusion criteria or meeting any of the above exclusion criteria
* Inability to safely participate in planned research (e.g., development of acute suicidal behavior during prior research participation)
* Unlikely to provide sufficient additional research data

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with schizophrenia-spectrum illness from the community.
Sampling Method: Non-Probability Sample
Enrollment: 648 (Actual)
Dates: Start 1989-09-15 (Actual)

PRIMARY OUTCOMES:
To map the physiological fMRI BOLD response, the brain electrical activity through MEG response and the blood flow, presynaptic and post-synaptic dopaminergic function through PET studies during different cognitive tasks | ongoing
  To map the physiological fMRI BOLD response, the brain electrical activity through MEG response and the blood flow, presynaptic and post-synaptic dopaminergic function through PET studies during different cognitive tasks
To explore the neuropsychological response in research subjects with schizophrenia under placebo conditions without the confounding effect of antipsychotics. | ongoing
  To explore the neuropsychological response in research subjects with schizophrenia under placebo conditions without the confounding effect of antipsychotics.

SECONDARY OUTCOMES:
PANSS data will be collected to determine changes or lack thereof in clinical status during the protocol. | Ongoing
  PANSS data will be collected to determine changes or lack thereof in clinical status during the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel P Eisenberg, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Because a large share of the accrued dataset precludes broad sharing language in the consent, it is unlikely that sharing of only some IPD that underlie results in any given publication would be of scientific value.

REFERENCES:
- [Background] Egan MF, Goldberg TE, Kolachana BS, Callicott JH, Mazzanti CM, Straub RE, Goldman D, Weinberger DR. Effect of COMT Val108/158 Met genotype on frontal lobe function and risk for schizophrenia. Proc Natl Acad Sci U S A. 2001 Jun 5;98(12):6917-22. doi: 10.1073/pnas.111134598. Epub 2001 May 29. PMID 11381111
- [Background] Meyer-Lindenberg A, Miletich RS, Kohn PD, Esposito G, Carson RE, Quarantelli M, Weinberger DR, Berman KF. Reduced prefrontal activity predicts exaggerated striatal dopaminergic function in schizophrenia. Nat Neurosci. 2002 Mar;5(3):267-71. doi: 10.1038/nn804. PMID 11865311
- [Derived] Rubinstein DY, Eisenberg DP, Carver FW, Holroyd T, Apud JA, Coppola R, Berman KF. Spatiotemporal Alterations in Working Memory-Related Beta Band Neuromagnetic Activity of Patients With Schizophrenia On and Off Antipsychotic Medication: Investigation With MEG. Schizophr Bull. 2023 May 3;49(3):669-678. doi: 10.1093/schbul/sbac178. PMID 36772948
- [Derived] Eisenberg DP, Kohn PD, Hegarty CE, Smith NR, Grogans SE, Czarapata JB, Gregory MD, Apud JA, Berman KF. Clinical correlation but no elevation of striatal dopamine synthesis capacity in two independent cohorts of medication-free individuals with schizophrenia. Mol Psychiatry. 2022 Feb;27(2):1241-1247. doi: 10.1038/s41380-021-01337-1. Epub 2021 Nov 17. PMID 34789848
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1989-M-0160.html